CLINICAL TRIAL: NCT00109746
Title: A Novel Therapy for Glucose Intolerance in HIV Disease
Brief Title: Use of a Nutritional Supplement to Treat Diabetic Symptoms in HIV-Infected Adults
Acronym: NT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Principal Investigator, Marie Gelato, Principal Investigator, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R21 AT002499-01A1
Record Dates: First submitted 2005-05-02; First posted 2005-05-03 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2013-05

CONDITIONS: Insulin Resistance; HIV Infections
Keywords: HIV; Treatment Experienced; Anti-Retroviral Agents; Antiretroviral Therapy, Highly Active; Picolinic acid; Dietary Supplements
MeSH Terms: conditions — Insulin Resistance; HIV Infections | interventions — picolinic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chromium Picolinate (Active Comparator): HIV+ and control may receive 500µg of chromium picolinate or placebo twice daily for two months.
  Interventions: Dietary Supplement: chromium picolinate
- Placebo (No Intervention): HIV+ and control may receive 500µg of chromium picolinate or placebo twice daily for two months.

INTERVENTIONS:
Dietary Supplement: chromium picolinate — HIV+ and control may receive 500µg of chromium picolinate or placebo twice daily for two months.
  Arms: Chromium Picolinate

SUMMARY:
The purpose of this study is to determine the effectiveness of the nutritional supplement chromium picolinate in improving insulin resistance, a symptom of diabetes, in HIV-infected patients. The ultimate goal is to find a simple therapy that can prevent the development of diabetes in individuals with HIV.

DETAILED DESCRIPTION:
Insulin resistance occurs when blood glucose levels get too high for the body to respond. Certain anti-HIV drugs are associated with increased insulin resistance and may lead to abnormal fat distribution, hypertension, and type 2 diabetes mellitus. The dietary supplement chromium picolinate has been shown to safely improve insulin sensitivity in patients with type 2 diabetes mellitus with no serious side effects. However, the effects of the supplement have not been thoroughly examined in HIV-infected individuals. This study will determine the effectiveness of chromium picolinate in improving insulin resistance in HIV-infected individuals.

This study will last 2 months. Participants will be randomly assigned to receive either chromium picolinate or placebo once a day for 2 months. Participants will have four overnight visits at the research center and two additional daytime visits for safety monitoring. During the overnight visits, participants will undergo a euglycemic hyperinsulinemic clamp, in which a continuous infusion of insulin is given through a vein and glucose levels are monitored through blood samples taken every 5 to 10 minutes. Fat tissue biopsies will also be conducted at the overnight study visits. During the safety monitoring visits, blood collection will occur for kidney and liver function tests, CD4 count, and viral load assessment.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Currently taking an anti-HIV drug regimen
* Insulin Resistant:fasting glucose between 5.56 and 7mmol/L and/or two hour post-glucose load between 7.78 and 11.11mmol/L

Exclusion Criteria:

* Cancer
* Acute illness that would interfere with the study
* Hypogonadism
* Hypothyroidism
* Untreated hypertension
* CD4 count less than 300 cells/mm3
* Viral load greater than 35,000 copies/ml
* Untreated hepatitis C virus infection
* Pregnancy
* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-11; Primary Completion 2009-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Improvement in insulin sensitivity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marie C. Gelato, MD, PhD, Principal Investigator — State University of New York/General Clinical Research Center
Locations (1):
- State University of New York/General Clinical Research Center, Stony Brook, New York, United States

REFERENCES:
- [Background] El-Sadr WM, Mullin CM, Carr A, Gibert C, Rappoport C, Visnegarwala F, Grunfeld C, Raghavan SS. Effects of HIV disease on lipid, glucose and insulin levels: results from a large antiretroviral-naive cohort. HIV Med. 2005 Mar;6(2):114-21. doi: 10.1111/j.1468-1293.2005.00273.x. PMID 15807717
- [Background] Howard AA, Floris-Moore M, Arnsten JH, Santoro N, Fleischer N, Lo Y, Schoenbaum EE. Disorders of glucose metabolism among HIV-infected women. Clin Infect Dis. 2005 May 15;40(10):1492-9. doi: 10.1086/429824. Epub 2005 Apr 11. PMID 15844072
- [Background] Taiwo BO. Insulin resistance, HIV infection, and anti-HIV therapies. AIDS Read. 2005 Apr;15(4):171-6, 179-80. PMID 15844237